CLINICAL TRIAL: NCT03378076
Title: A Randomized, Open-label, Parallel Group Study in Patients With Bilateral Knee Osteoarthritis Comparing the Systemic Exposure of Triamcinolone Acetonide Following Administration Into Both Knees of Either Extended-release FX006 or Immediate-release TAcs (Triamcinolone Acetonide Suspension)
Brief Title: Study to Compare Exposure of TA Following Administration of Either FX006 or TAcs in Patients With Bilateral Knee OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FX006-2017-012
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Results first posted 2019-05-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Bilateral Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Corticosteroid; Bilateral; Pain; Intra-articular; Injection
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — FX006; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FX006 32 mg (Experimental): Two intra-articular (IA) injections of FX006 32 mg (total dose of 64 mg)
  Interventions: Drug: FX006 32 mg
- TAcs 40 mg (Active Comparator): Two intra-articular (IA) injections of TAcs 40 mg (total dose of 80 mg)
  Interventions: Drug: TAcs 40 mg

INTERVENTIONS:
Drug: FX006 32 mg — Drug: Extended-release 32 mg FX006 IA injection into each knee (total 64 mg dose)
  Other Names: Zilretta
  Arms: FX006 32 mg
Drug: TAcs 40 mg — Drug: Immediate-release 40mg TAcs IA injection into each knee (total 80 mg dose)
  Other Names: Kenalog®-40 Injection; Triamcinolone Acetonide Crystalline Suspension (TAcs); TCA-IR 40
  Arms: TAcs 40 mg

SUMMARY:
This is a randomized, open-label, parallel group study to compare systemic exposure of triamcinolone acetonide following administration into both knees of either FX006 or TAcs.

DETAILED DESCRIPTION:
This is a randomized, open label, parallel group study that will be conducted in male and female patients ≥ 40 years of age with bilateral knee OA.

Approximately 24 patients will be randomized to one of two treatment groups (1:1) and treated with IA injections to both knees of either:

* extended-release FX006 64 mg total dose (approximately 12 patients) or
* immediate-release TAcs 80 mg total dose (approximately 12 patients) Each patient will be screened to confirm the diagnosis of OA and eligibility based on the inclusion/exclusion requirements and will be randomized to treatment on Day 1. Following screening, pharmacokinetics (PK) and safety will be evaluated at 6 out-patient visits scheduled on Study Days 1 [calendar day of injection], 2, 8, 15, 29, and 43.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Male or female greater than or equal to 40 years of age
* Symptoms consistent with OA in both knees for greater than or equal to 6 months prior to Screening (patient reported is acceptable)
* Currently meets ACR Criteria (clinical and radiological) for OA in both knees
* Knee pain in both knees for greater than 15 days over the last month (as reported by the patient)
* Body mass index (BMI) less than or equal to 40 kg/m2
* Morning serum cortisol result within normal range at Screening (5-23 mcg/dL or 138-635 nmol/dL)
* Ambulatory and in good general health
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions.
* Willing to abstain from use of protocol-restricted medications during the study

Exclusion Criteria:

* Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* History of infection in either knee joint
* Clinical signs and symptoms of active knee infection or crystal disease in either knee within 1 month of Screening
* Unstable joint (such as a torn anterior cruciate ligament) in either knee within 12 months of Screening
* Presence of surgical hardware or other foreign body in either knee
* Surgery or arthroscopy of either knee within 12 months of Screening
* IA treatment of any joint with any of the following agents within six (6) months of Screening: any corticosteroid preparation (investigational or marketed, including FX006), any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection; investigational or marketed).
* IA treatment in either knee with hyaluronic acid (investigational or marketed) within 6 months of Screening
* Parenteral or oral corticosteroids (investigational or marketed) within 3 months of Screening
* Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening
* Females who are pregnant or nursing or plan to become pregnant during the study; men who plan to conceive during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (3):
- United States (3):
  - LA Biomed at Harbor-UCLA Medical Center, Torrance, California
  - Rochester Clinical Research, Rochester, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

REFERENCES:
- [Derived] Kivitz A, Kwong L, Shlotzhauer T, Lufkin J, Cinar A, Kelley S. A randomized, phase IIa study to assess the systemic exposure of triamcinolone acetonide following injection of extended-release triamcinolone acetonide or traditional triamcinolone acetonide into both knees of patients with bilateral knee osteoarthritis. Ther Adv Musculoskelet Dis. 2019 Oct 16;11:1759720X19881309. doi: 10.1177/1759720X19881309. eCollection 2019. PMID 31662801

RESULTS

PARTICIPANT FLOW:
Groups:
- FX006 32 mg: 12 subjects received FX006 32 mg as a single 5 mL IA injection into each knee for a total of total 64 mg dose
- TAcs IR 40 mg: 12 subjects received TAcs 40 mg as a single 5 mL IA injection into each knee for a total 80 mg dose
Period: Overall Study
Arm/Group | FX006 32 mg | TAcs IR 40 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FX006 64 mg; TAcs IR 80mg: Single 5 mL IA injection into each knee
- Total: Total of all reporting groups
Arm/Group | FX006 64 mg | TAcs IR 80mg | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (6.45) | 61.6 (8.17) | 61.7 (7.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.31 (3.669) | 30.35 (4.955) | 31.83 (4.524)

OUTCOME MEASURES:

1. Primary Outcome: Measure the Concentration of Triamcinolone Acetonide (TA) in Blood Plasma
Description: Plasma drug concentrations (pg/mL) by Time Point across FX006 and TAcs treatment arms in plasma.
  For the PK analysis and individual concentration vs. time plots, a concentration that is BLOQ is assigned a value of zero if it occurs in a profile before the first measurable concentration. If a BLOQ value occurs after a measurable concentration in a profile and is followed by a value above the lower limit of quantification, then the BLOQ is treated as missing data. If a BLOQ value occurs at the end of the collection interval (after the last quantifiable concentration) it is set to zero. If two BLOQ values occur in succession after Cmax, the profile is deemed to have terminated at the first BLOQ value and any subsequent concentrations are set to zero for PK calculations
Time Frame: 43 days
Population: All patients who received 2 IA injections (one in each knee) of study drug, completed scheduled sampling, and had sufficient plasma concentration data
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- FX006 32 mg: Two 5 mL IA injections (total dose of 64 mg)
- TAcs 40 mg: Two 1mL IA injections (total dose of 80 mg)
Arm/Group | FX006 32 mg | TAcs 40 mg
Number analyzed (Participants) | 12 | 12
pg/mL
  Day 1- Hour 1 | 1801.5 [1261.50 to 2572.77] | 4507.9 [1205.43 to 16857.74]
  Day 1 - Hour 2 | 1893.6 [1328.58 to 2698.84] | 5140.1 [1327.67 to 19899.79]
  Day 1 - Hour 3 | 1958.1 [1336.54 to 2868.86] | 5443.8 [1357.81 to 21825.90]
  Day 1 - Hour 4 | 2013.8 [1381.39 to 2935.59] | 5454.2 [1409.98 to 21098.36]
  Day 1 - Hour 5 | 1914.4 [1291.93 to 2836.82] | 5338.9 [1366.93 to 20852.59]
  Day 1 - Hour 6 | 1900.2 [1293.77 to 2790.96] | 5430.6 [1442.24 to 20448.57]
  Day 1 - Hour 8 | 1928.1 [1288.45 to 2885.17] | 5199.0 [1418.52 to 19054.80]
  Day 1 - Hour 10 | 1839.8 [1241.72 to 2725.96] | 4948.8 [1392.07 to 17593.31]
  Day 1 - Hour 12 | 1793.9 [1247.06 to 2580.66] | 4507.8 [1294.51 to 15697.14]
  Day 2 - Hour 24 | 1948.8 [1349.93 to 2813.36] | 4185.4 [1614.39 to 10850.75]
  Day 8 | 1397.0 [1073.13 to 1818.65] | 450.8 [230.66 to 880.92]
  Day 15 | 956.2 [759.23 to 1204.25] | 428.7 [231.92 to 792.29]
  Day 29 | 445.8 [313.12 to 634.80] | 334.6 [182.45 to 613.80]
  Day 43 | 265.8 [199.56 to 354.03] | 241.0 [119.11 to 487.54]

2. Primary Outcome: Incidence of Treatment Emergent Adverse Events
Description: Safety analyses were conducted using the safety population.
  Analyses of adverse events will be performed for those events that are considered treatment emergent, where treatment emergent is defined as any adverse event with onset after the administration of study medication in the first knee through the end of the study or any event that was present at baseline but worsened in intensity through the end of the study. Severity of Adverse events were graded by the Principal Investigator using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The grading went from Grade 1 (Mild) to Grade 5 (Death related to AE).
Time Frame: 43 days
Population: All patients who received study drug (injection in at least one knee).
Measure: Number; unit: participants
Arm/Group | FX006 32 mg | TAcs 40 mg
Number analyzed (Participants) | 12 | 12
participants
  Patients with TEAE Grade 1 | 6 | 3
  Patients with TEAE Grade 2 | 1 | 2
  Patients with TEAE Grade 3 | 1 | 0
  Patients with TEAE Grade 4 | 0 | 0
  Patients with TEAE Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following IA administration through the final study visit at 43 days.
Groups:
- FX006 32 mg: Two 5 mL intra-articular injection
  FX006: Sustained Release Steroid
- TAcs 40 mg: Commercially available triamcinolone acetonide, two 1 mL intra-articular injection
  TAcs: Immediate Release Steroid
Arm/Group | FX006 32 mg | TAcs 40 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg (N=12) | TAcs 40 mg (N=12)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection Site Pain (General disorders) | 1 (1) | 0 (0)
Vessel Puncture Site Haematoma (General disorders) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03378076/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03378076/SAP_001.pdf